CLINICAL TRIAL: NCT00164606
Title: A Dissemination Trial of the Positive Parenting Program to Reduce Child Maltreatment in South Carolina
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Centers for Disease Control and Prevention (U.S. Federal Agency)
Allocation: Randomized | Model: Factorial | Purpose: Prevention
Other Study IDs: CDC-NCIPC-3838; U17/CCU422317-01
Record Dates: First submitted 2005-09-12; First posted 2005-09-14 (Estimated); Last update posted 2007-09-21 (Estimated); Status verified 2007-09

CONDITIONS: Child Abuse
Keywords: child maltreatment; child abuse; prevention

INTERVENTIONS:
Behavioral: Positive Parenting Program (Triple-P)

SUMMARY:
This is a population-based evaluation of the effectiveness of the Triple-P-Positive Parenting Program. Triple-P is a system of parenting programs with multiple levels that aims to provide parents with parenting skills and support.

DETAILED DESCRIPTION:
Eighteen counties in the state of South Carolina will be randomized to the dissemination of the Triple-P system or to a waitlist control condition. University of South Carolina staff will train health care professionals in the nine dissemination counties to use the Triple-P parenting programs. Triple-P is a parenting program that uses a tiered system of interventions of increasing strength depending on parents' and children's differing needs, ranging from media and information-based strategies, to two levels of moderate-intensity intervention using a brief consultation format, to two more intensive levels of parent training and behavioral family intervention targeting parenting skills and other family adversity factors such as marital conflict, depression and high levels of parenting stress. The evaluation of the dissemination of Triple-P will rely on two methods: the analysis of aggregate data on child maltreatment, injuries and hospitalizations, and annual surveys of families to examining parenting education, practices, and child behavior.

ELIGIBILITY:
Inclusion Criteria:

* Counties in South Carolina

Max Age: 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 14690 (Estimated)
Dates: Start 2003-05; Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
child maltreatment reports
injury to children

CONTACTS AND LOCATIONS:
Overall Officials: Ronald J Prinz, PhD, Principal Investigator — University of South Carolina
Locations (1):
- University of South Carolina, Columbia, South Carolina, United States